CLINICAL TRIAL: NCT02562872
Title: Proof-of-concept, Single Center Study in Healthy Adult Volunteers to Investigate Safety, Tolerability, Pharmacokinetics and Prophylactic Activity of Single Dose DSM265 in a Controlled Human Malarial Infection Challenge Either by Direct Venous Inoculation of Plasmodium Falciparum Sporozoites or Mosquito-borne Plasmodium Falciparum
Brief Title: DSM265 Prophylaxis of Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); United States Department of Defense (U.S. Federal Agency); Center for Infectious Disease Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMV_DSM265_14_03; CDMRP-PR130402 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: Controlled; Human; Malaria; Infection; Healthy; Volunteer
MeSH Terms: conditions — Malaria; Infections | interventions — DSM265; Sporozoites

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 Active DSM265 (Experimental)
  Interventions: Drug: DSM265; Biological: Sporozoites
- Cohort 1 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Biological: Sporozoites
- Cohort 2a Active DSM265 (Experimental)
  Interventions: Drug: DSM265; Biological: Sporozoites
- Cohort 2a Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Biological: Sporozoites
- Cohort 2b Active DSM265 (Experimental)
  Interventions: Drug: DSM265; Biological: Infective mosquito bite
- Cohort 2b Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Biological: Infective mosquito bite

INTERVENTIONS:
Drug: DSM265 — DSM265 400 mg single oral dose
  Arms: Cohort 1 Active DSM265; Cohort 2a Active DSM265; Cohort 2b Active DSM265
Drug: Placebo — Placebo to match DSM265, single oral dose
  Arms: Cohort 1 Placebo; Cohort 2a Placebo; Cohort 2b Placebo
Biological: Sporozoites — Direct venous inoculation of 3200 cryopreserved Plasmodium falciparum (NF54 strain) sporozoites
  Other Names: PfSPZ
  Arms: Cohort 1 Active DSM265; Cohort 1 Placebo; Cohort 2a Active DSM265; Cohort 2a Placebo
Biological: Infective mosquito bite — Five single bites by laboratory reared female Anopheles stephensi mosquitoes carrying Plasmodium falciparum
  Arms: Cohort 2b Active DSM265; Cohort 2b Placebo

SUMMARY:
The study is a single centre, randomised, placebo-controlled, double-blind study with DSM265 including up to two cohorts of healthy male and female volunteers aged 18 to 45 years.

The study will be conducted into two sequential parts (Cohort 1 and Cohorts 2a and 2b).

DETAILED DESCRIPTION:
Cohort 1:

* Controlled human malaria infection on Day 0 (Direct Venous Inoculation of 3200 cryopreserved Plasmodium falciparum sporozoites)
* Drug administration on Day -3
* 8 subjects: 6 DSM265 400 mg: 2 matching placebo Clinical safety review of Cohort 1 in order to proceed to Cohorts 2a and 2b

Cohort 2a:

* Controlled human malaria infection on Day 0 (Direct Venous Inoculation of 3200 cryopreserved Plasmodium falciparum sporozoites)
* Drug administration on Day -X (to be defined following safety and pharmacokinetic data)
* 8 subjects: 6 DSM265 400 mg: 2 matching placebo

Cohort 2b:

* Controlled human malaria infection on Day 0 (infected mosquito bite)
* Drug administration on Day -X (to be defined following safety and pharmacokinetic data)
* 8 subjects: 6 DSM265 400 mg: 2 matching placebo

ELIGIBILITY:
* Good health based on medical history and physical examination
* body mass index >18 and <30kg/m2
* Laboratory results without clinically significant findings within 60 days
* Males must use medically acceptable form of contraception from the dose of DSM265/Placebo for 120 days
* Women must be of non-child bearing potential or willing and able to practice one of the required continuous acceptable methods of contraception and have negative pregnancy tests
* Able & willing to comply with all study requirements throughout the study
* Agree to undergo all study procedures, attend all study visits and stay overnight for observation if required, to last follow-up visit
* Willing to undergo a controlled human malaria infection by mosquito bites / inoculation
* Able and willing to answer all questions on informed consent correctly, and to sign the informed consent form
* Reachable constantly by mobile phone or email throughout the study period
* Refrain from blood donation throughout the study
* Willing to take atovaquone-proguanil, Chloroquine or other registered antimalarial

Exclusion Criteria:

* Any history of malaria; any severe reactions to mosquito or insect bites; any history of anaphylaxis
* Plans to travel to malaria endemic region during the study period
* Previous participation in any malaria vaccine study or controlled human malaria infection study
* Participation in any other clinical study within 30 days of enrollment or plan to participate in another investigational vaccine/drug research during the study
* Breastfeeding or planning to become pregnant during the time of the study
* Positive Human Immunodeficiency Virus, Hepatitis B or C tests
* Any confirmed/suspected immunosuppressive or immunodeficient state
* History of serious psychiatric condition that may affect participation in the study, or history of convulsions, seizures, or of severe head trauma
* Symptoms, physical signs or laboratory values suggestive of systemic disorders
* History of cancer (except basal cell carcinoma of the skin)
* History of arrhythmias or documented prolonged QTcF-interval (>450 msec) or 12-lead ECG demonstrating specific abnormalities
* Moderate risk or higher for cardiovascular event within 5 years (>10%)
* Positive family history in 1st or 2nd degree relative <50 years for cardiac disease, or history of, or known active cardiac disease
* history of: psoriasis or porphyria which may be exacerbated by chloroquine; splenectomy, or sickle cell anaemia or other red blood cell disorders; allergy or contra-indication to chloroquine or atovaquone-proguanil
* Treatment with an investigational drug within 28 days or 5 half-lives of study medication; use of any drugs or dietary supplements within 7 days or 5 half-lives prior to study medication. Herbal supplements must be discontinued at least 28 days prior to study medication. As an exception, acetaminophen or ibuprofen may be used as approved by the investigator
* Use of any prohibited medication
* Grapefruit or product containing grapefruit from28 days before study medication or throughout the study
* History of drug or alcohol abuse within 12 months prior to dosing, or laboratory evidence of abuse
* Current smoking of more than 10 cigarettes or equivalent per day
* Plan for major surgery between enrolment and study completion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with positive parasitemia | 28 days
  positive parasitemia detected by qRT-PCR
Time interval between challenge and the first positive parasitemia | 28 days
  Time from infection to peripheral parasitemia (qRT-PCR) in DSM265 / placebo treated subjects in each cohort given as a geometric mean [days]

CONTACTS AND LOCATIONS:
Overall Officials: James G Kublin, MD/MPH, Principal Investigator — Fred Hutchinson Cancer Research Centre
Locations (1):
- Fred Hutchinson Cancer Research Center - Prevention Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No